CLINICAL TRIAL: NCT04179201
Title: Study on Prevalence, Risk Factors and Intestinal Microecology of Clostridium Difficile Infection in Chinese Patients With Inflammatory Bowel Disease
Brief Title: Study on Clostridium Difficile Infection in Chinese Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChiECRCT20190106
Record Dates: First submitted 2019-11-22; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Bowel Diseases; Clostridium Infections
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collecting stool samples from subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD with CDI: Inflammatory bowel disease with clostridium difficile infection
- IBD without CDI: Inflammatory bowel disease without clostridium difficile infection

SUMMARY:
In recent years, the incidence of Inflammatory Bowel Disease (IBD) has been increasing in China, which poses great challenges and burdens to the medical community due to its unknown etiology, recurrence and incurability. Co-infection is one of the important causes in IBD development. IBD accompanied with Clostridium Difficile Infection (CDI) can significantly decrease the treatment efficiency, leading to increased surgical rate, increased mortality, prolonged hospital stay, and increased hospital costs. Recently, several Chinese clinical guidelines about IBD or CDI have been published, but these guidelines are mainly based on the foreign studies. Compared with the developed countries, the lack of multi-center, large-scale and multi-test clinical trials and cohort studies caused limited understanding for IBD-CDI in China. Therefore, it is of great importance to carry out the multi-center clinical trials and analysis on IBD-CDI to improve the diagnostic and therapeutic efficiency in IBD-CDI patients

Objective:

1. To evaluate the prevalence rate of IBD-CDI in Chinese adults in China based on the multi-center clinical trials..
2. To analyze the related risk factors of IBD-CDI in China based on the multi-center clinical trials.
3. To analyze the intestinal flora of IBD-CDI patients via high-throughput sequencing.

ELIGIBILITY:
Inclusion Criteria:

* 1.Inpatients with diagnostic criteria for ulcerative colitis and Crohn's disease in accordance with the consensus opinion on the diagnosis and treatment of inflammatory bowel disease in China in 2012
* 2.Willing to participate in the study;
* 3. Have the ability to understand and sign informed consent.

Exclusion Criteria:

* 1.Patients with infectious enteritis, intestinal tuberculosis, lymphoma, Behcet's disease or other intestinal diseases except inflammatory bowel disease;
* 2.Pregnant or lactating women;
* 3.Severe circulatory system, respiratory system, blood system, immune system, urinary system and other combined diseases or serious psychosomatic diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population will be selected from six hospital in China.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence rate of IBD with CDI in Chinese adults | 3 years
  To analyze the prevalence rate of IBD with CDI in Chinese adults based on the multicenter clinical trials.

SECONDARY OUTCOMES:
Risk factors of IBD with CDI in China | 3 years
  To analyze the related risk factors of IBD with CDI in China based on the multicenter clinical trials. Including demographic data,severity of disease（Mayo score for ulcerative colitis and CDAI score for CD),laboratory results（ESR、CRP、WBC、Hb、RBC）and combination therapy.
Gut microbiota in patients with IBD-CDI，IBD and healthy volunteers by 16S rDNA sequencing | 3 years
  To analyze the gut microbiota with IBD-CDI，IBD and healthy volunteers.Including fecal flora composition and the abundance analysis by 16S rDNA sequencing.

OTHER OUTCOMES:
Using PCR and ELISA to detect the positive rate of clostridium difficile in patients with IBD and healthy volunteers | 3 years
  To compare the positive rate of clostridium difficile in patients with IBD and healthy volunteers by PCR and ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, PhD, Principal Investigator — Chief Professor of Xijing Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Xijing Hospital, Xi'an, Shaanxi
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Renji Hospital, Shanghai